CLINICAL TRIAL: NCT04728243
Title: WHO QualityRights Online Training for Mental Health Workers in Ghana
Brief Title: WHO QualityRights E-training in Ghana
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Society of Ghana (Other)
Collaborators: University of Cagliari (Other); Columbia University (Other); World Health Organization (Other); Mental Health Authority of Ghana (Unknown)
Responsible Party: Principal Investigator, Maria Francesca Moro, Principal Investigator and Researcher, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2021_1
Record Dates: First submitted 2021-01-20; First posted 2021-01-28 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Knowledge; Attitudes; Practices
Keywords: mental health; human rights; RCT; Ghana; online training
MeSH Terms: conditions — Behavior; Psychological Well-Being

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WHO QualityRights (Experimental): Mental health professionals assigned to the experimental arm will be enrolled in the WHO QualityRights online training.
  Interventions: Other: WHO QualityRights e-training
- WHO Coronavirus Disease of 2019 (COVID19) (Placebo Comparator): Mental health professionals assigned to the control arm will be enrolled in the WHO novel coronavirus 2019 online training series.
  Interventions: Other: WHO COVID-19 online training

INTERVENTIONS:
Other: WHO QualityRights e-training — The WHO QualityRights online training aims to increase knowledge about the rights of people with psychosocial disabilities and change negative attitudes towards these persons and their role as rights holders. Furthermore, the training provides mental health professionals with the skills necessary to support people with psychosocial disabilities to advocate for their rights. The WHO QualityRights online training includes five core modules: 1) Human rights; 2) Mental health, disability, and human rights; 3) The right to health and recovery; 4) Legal capacity and the right to decide; 5) Free from coercion, violence, and abuse. Each module is composed of presentations, videos, interactive exercises, and forum discussions involving all participants. In the online training forum discussions, particular attention will be given to issues relevant to the Ghanaian context.
  Arms: WHO QualityRights
Other: WHO COVID-19 online training — The WHO novel coronavirus 2019 online training series provides a general introduction to COVID-19 and similar respiratory infections and information on what facilities and professionals should be doing to prevent and respond to COVID-19 cases. The training is similar in length to the WHO QualityRights training (13 h 15 min vs. 19 hours) and is intended for health professionals and other stakeholders.
  Arms: WHO Coronavirus Disease of 2019 (COVID19)

SUMMARY:
This is a cluster randomized controlled trial to determine the efficacy of the WHO QR online training compared with a placebo intervention in improving the knowledge about human rights, the attitudes towards people with psychosocial disabilities, and the practices related to substitute-decision making and coercion among mental health professionals.

Given the impact human rights violations have on the health of persons with psychosocial disabilities, an effort is needed to carry out methodologically strong research in this area. The study proposed will provide robust evidence to support further investment in interventions such as the WHO QualityRights training and make steps forward promoting the rights of people with psychosocial disabilities.

DETAILED DESCRIPTION:
Background. People with psychosocial disabilities are commonly exposed to human rights violations within the mental health care system and in the general community. Such violations occur in all countries and are not only a problem from an ethical point of view but additionally have profound repercussions on the health of persons with psychosocial disabilities. Although psychiatric facilities are the very institutions responsible for the care and support of people with psychosocial disabilities, they are also often places in which persons with psychosocial disabilities are victims of inhumane treatments, including psychological, physical, and sexual abuse or violence. To stop these human rights violations, there is a need to reform mental health systems and thus change mental health professionals' practices leading to violations of people with psychosocial disabilities' rights. However, for this to happen, two main barriers need to be addressed. One barrier is the lack of human rights literacy among mental health professionals. The second barrier is that many mental health professionals hold negative attitudes towards people with psychosocial disabilities.

Recently, the World Health Organization (WHO) has developed the QualityRights (QR) online training. This training includes modules to increase knowledge about the rights of people with psychosocial disabilities and change the negative attitudes towards them and their role as rights holders. Furthermore, the training provides mental health providers with the skills necessary to advocate for a human rights-based approach in mental health. Currently, there is a growing interest in the QualityRights training, and the WHO is implementing it in different countries. However, the efficacy of this intervention has not been rigorously evaluated.

Objectives. To determine the efficacy of the QR online training compared with a placebo intervention (online training on Coronavirus Disease - 2019) in improving the knowledge about human rights, the attitudes towards people with psychosocial disabilities, and the practices related to substitute-decision making and coercion among mental health professionals.

Methods. This is a cluster randomized controlled trial (cRCT) being conducted in Ghana. An estimated sample of 252 mental health professionals will be recruited from across 28 clusters within three psychiatric hospitals. Participants will be divided in two arms to receive either the WHO QR online training on human rights issues in mental health or the WHO Coronavirus online training for health professionals. The primary outcomes, assessed post-training, at 3 months, and at 6 months are increase in the knowledge about human rights and mental health and improvement on the attitudes towards persons with psychosocial disabilities. Secondary outcomes, assessed at 3 and 6 months, consist of improvements in the mental health professionals' practices, burn-out levels, and well-being. All data will be collected online.

Discussion. Given the impact human rights violations have on the health of persons with psychosocial disabilities, an effort is needed to carry out methodologically strong research in this area. The study proposed will provide robust evidence to support further investment in interventions such as the WHO QualityRights training and make steps forward promoting the rights of people with psychosocial disabilities.

ELIGIBILITY:
Inclusion Criteria:

* Able to speak English. English is an official language of Ghana and is used as a lingua franca throughout the country. English is also the most used of the eleven official languages spoken in Ghana .
* Mental health professionals currently working in the in-patient units of the three psychiatric hospitals selected for the study (all in the Accra area)

Exclusion Criteria:

* Persons who participated to the in-person WHO QualityRights trainings held in Ghana.
* Persons enrolled in the online WHO QualityRights training. .

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2023-01-19 (Actual)

PRIMARY OUTCOMES:
Change from Baseline knowledge about human rights of persons with psychosocial disabilities post-training | pre-training, immediately post-training
  World Health Organization's Knowledge about the Rights of persons with psychosocial disabilities questionnaire: Questionnaire to assess knowledge about the rights included in the United Nations Convention on the Rights of Persons with Disabilities. Scores range between 0 and 23. Higher score indicates higher level of knowledge.
Change from Baseline attitudes towards persons with psychosocial disabilities role as rights-holders post-training | pre-training, immediately post-training
  World Health Organization's questionnaire on the attitudes towards people with psychosocial disabilities as rights-holders. Scores range between 17 and 85. Higher score indicates more negative attitudes.

SECONDARY OUTCOMES:
Change from Baseline Practices related to substitute-decision making and coercion scale at 3 months | pre-training, at 3 months
  Practices related to substitute-decision making and coercion questionnaire. Scale to measure the use of substitute-decision making and coercive practices in mental health units. This questionnaire includes two sub-scales. The first range is between 7 and 49. A high score indicates practices related to substitute-decision making and coercion are used frequently by the respondent. The second range is between 5 and 25. High scores indicate that the mental health professionals working in the units of the respondents are more willing to use practices related to substitute-decision making and coercion than they are.
Change from Baseline Seclusion and Restraint Experience post-training | pre-training, immediately post-training
  Seclusion and Restraint Experience Questionnaire (SREQ) - modified version. Questionnaire to measure emotional and ethical experiences linked to the use of seclusion and restraint among health professionals. Scores range between 25 and 100. Higher scores indicates higher endorsement of specific experiences.
Change from Baseline Burnout at 3 months | pre-training, at 3 months
  Abbreviated Maslach Burnout Inventory (MBI). Inventory to measure burn-out among health professionals. Scores range between 9 and 27. Higher scores indicate higher burnout.
Change from Baseline Quality of Life at 3 months | pre-training, at 3 months
  World Health Organization Quality of Life (WHOQOL-BREF)Questionnaire to measure quality of life during the last month. Scores range between 0 and 100. Higher scores denote higher quality of life.

OTHER OUTCOMES:
Change from Baseline knowledge about human rights of persons with psychosocial disabilities at 3 months | pre-training, at 3 months
  World Health Organization's Knowledge about the Rights of persons with psychosocial disabilities questionnaire: Questionnaire to assess knowledge about the rights included in the United Nations Convention on the Rights of Persons with Disabilities. Scores range between 0 and 23. Higher score indicates higher level of knowledge.
Change from Baseline knowledge about human rights of persons with psychosocial disabilities at 6 months | pre-training, at 6 months
  World Health Organization's Knowledge about the Rights of persons with psychosocial disabilities questionnaire: Questionnaire to assess knowledge about the rights included in the United Nations Convention on the Rights of Persons with Disabilities. Scores range between 0 and 23. Higher score indicates higher level of knowledge.
Change from Baseline attitudes towards persons with psychosocial disabilities role as rights-holders at 3 months | pre-training, at 3 months
  World Health Organization's questionnaire on the attitudes towards people with psychosocial disabilities as rights-holders. Scores range between 17 and 85. Higher score indicates more negative attitudes.
Change from Baseline attitudes towards persons with psychosocial disabilities role as rights-holders at 6 months | pre-training, at 6 months
  World Health Organization's questionnaire on the attitudes towards people with psychosocial disabilities as rights-holders. Scores range between 17 and 85. Higher score indicates more negative attitudes.
Change from Baseline Practices related to substitute-decision making and coercion scale at 6 months | pre-training, at 6 months
  Scale to measure the use of substitute-decision making and coercive practices in mental health units. This questionnaire includes two sub-scales. The first range is between 7 and 49. A high score indicates practices related to substitute-decision making and coercion are used frequently by the respondent. The second range is between 5 and 25. High scores indicate that the mental health professionals working in the units of the respondents are more willing to use practices related to substitute-decision making and coercion than they are.
Change from Baseline Burnout at 6 months | pre-training, at 6 months
  Abbreviated Maslach Burnout Inventory (MBI). Inventory to measure burn-out among health professionals. Scores range between 9 and 27. Higher scores indicate higher burnout.
Change from Baseline Quality of Life at 6 months | pre-training, at 6 months
  World Health Organization Quality of Life (WHOQOL-BREF) Questionnaire to measure quality of life during the last month. Scores range between 0 and 100. Higher scores denote higher quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Maria Francesca Moro, M.D., Principal Investigator — Columbia University
Locations (3):
- Ghana (3):
  - Ankaful Psychiatric Hospital, Cape Coast, Central Region
  - Accra Psychiatric Hospital, Accra
  - Pantang Psychiatric Hospital, Accra

IPD SHARING:
Plan to Share IPD: Yes
A coded dataset, with no confidential information, will be shared with researchers at Columbia University for data analysis collaboration
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: to be decided
Access Criteria: to be decided - the access criteria will guarantee the respect of confidentiality in agreement with General Data Protection Regulation (GDPR) and HIPAA requirements

REFERENCES:
- [Derived] Moro MF, Gyimah L, Susser E, Ansong J, Kane JC, Osei A, Gureje O, Kofie H, Taylor D, Drew N, Ohene SA, Fatawu A, Addico NL, Atzeni M, D'Oca S, Funk M, Carta MG. Evaluating the efficacy of the WHO QualityRights e-training in promoting the rights of persons with mental health conditions and psychosocial disabilities: a cluster randomised controlled trial in Ghana. BMJ Glob Health. 2025 Dec 9;10(12):e021215. doi: 10.1136/bmjgh-2025-021215. PMID 41365627